CLINICAL TRIAL: NCT05672901
Title: Comparison of a Novel Silicone Gel Vs. Estrogen Vaginal Cream for the Management of Genitourinary Syndrome of Menopause: a Non-inferiority Trial
Brief Title: Silicone Gel Vs. Estrogen Vaginal Cream for the Management of Genitourinary Syndrome of Menopause
Acronym: VITAL-E
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stratpharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPAMG02
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Genitourinary Syndrome of Menopause
MeSH Terms: interventions — Estradiol; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- StrataMGT (Experimental): Participants will apply StrataMGT (silicone gel) 2-5 times daily (no limit in application times) to treat GSM for 3 months.
  Interventions: Device: StrataMGT
- Estrace (Active Comparator): Participants will receive Estrace vaginal cream (estrogen) to treat GSM for 3 months. Application will be 1 g daily for the first two weeks. Afterwards, a maintenance dosage of 1 g three times a week is applied.
  Interventions: Drug: Estrace 0.01% Vaginal Cream

INTERVENTIONS:
Device: StrataMGT — StrataMGT is a 100% medical grade film-forming silicone gel for the treatment of cutaneous skin lesions and Genitourinary Syndrome of Menopause. StrataMGT is a flexible wound dressing used on compromised skin. It dries to form a thin, flexible wound dressing which hydrates and protects affected areas. StrataMGT is used to relieve low grade inflammatory changes such as dry, itching, flaking, peeling and irritated skin. StrataMGT is designed for partially epithelized skin and is suitable for children and patients with sensitive skin.
  Arms: StrataMGT
Drug: Estrace 0.01% Vaginal Cream — Estrace is a prescriptive female hormone indicated in the treatment of moderate to severe symptoms of Genitourinary Syndrome of Menopause.
  Arms: Estrace

SUMMARY:
The goal of this randomized controlled trial is to test the efficacy of StrataMGT in the management of Genitourinary Syndrome of Menopause (GSM) compared to estrogen therapy. The main question it aims to answer is:

- Will StrataMGT be non-inferior regarding patient quality of life compared to standard of care?

Participants will use either StrataMGT or estrogen vaginal cream to treat GSM for 3 consecutive months. After the baseline assessment, participants will be assessed monthly for quality of life, clinical signs, symptoms, pathology and adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Confirmed postmenopausal age
* Diagnosed genitourinary syndrome of menopause
* Access to a smartphone, tablet or computer, and to a functional email address.

Exclusion Criteria:

* Contraindication for the use of estrogen therapy
* Unable to provide informed consent
* Patient unable to apply topical device
* Allergy or intolerance to ingredients or excipients of the formulation of studied products

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
PROM: Quality of Life | 3 months
  The improvement of patient quality of life will be assessed at baseline and during each monthly follow-up using the patient-rated Vulvar Disease Quality of Life (VQLI) Index questionnaire. Questions are rated on a numeric scale from 0 (not at all) - 3 (very much). This outcome is patient-rated, thus unblinded.

SECONDARY OUTCOMES:
Clinical signs | 3 months
  Signs are rated by the investigator (blinded) during baseline and at the final visit after 3 months, using a combination of visual assessment and categorical scale ranging from 0=normal to 10=worst possible.
Adverse Reactions | 3 months
  Adverse reactions are rated by the investigator (blinded) during baseline and at the final visit after 3 months, using a combination of visual assessment and categorical scale ranging from 0=normal to 10=worst possible.
Visual pathology | 3 months
  Severity of the visual pathology is rated by the investigator (blinded) during baseline and at the final visit after 3 months, using a combination of visual assessment and categorical scale ranging from 0=normal to 10=worst possible.
PROM: Symptoms | 3 months
  Symptoms are rated by the patient at baseline and during each monthly follow-up, using a combination of visual assessment and categorical scale ranging from 0=normal to 10=worst possible. This outcome is patient-rated, thus unblinded.
PROM: Dyspareunia | 3 months
  Dyspareunia is rated by the patient at baseline and during each monthly follow-up, using a combination of visual assessment and categorical scale ranging from 0=normal to 10=worst possible. This outcome is patient-rated, thus unblinded.
PROM: Product Rating | 3 months
  Product performance is rated by the patient at the final visit after 3 months, using a Likert scale from 1=unsatisfactory to 5=excellent. This outcome is patient-rated, thus unblinded.
PROM: Treatment Adherence | 3 months
  Treatment adherence is reported by the patient during the final study assessment, indicating the number of days/week and times/day the product was applied during the previous month. Percentage of treatment adherence is calculated from the minimum required treatment schedule.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Orange Coast Women's Medical Group, Laguna Hills, California
  - Abba Medical Group, Miami, Florida
  - One Health Research Clinic, Johns Creek, Georgia

IPD SHARING:
Plan to Share IPD: No